CLINICAL TRIAL: NCT06072378
Title: The Computational and Neural Mechanisms Linking Decision-making and Memory in Humans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Salman Ehtesham Qasim, Ph.D., Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro2024002100; K99MH132873 (NIH)
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Memory, Short-Term

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Value-manipulation (Experimental): Participants with epilepsy will complete a behavioral task in which they use a laptop computer to do a decision-making and memory task.
  Interventions: Behavioral: Value-manipulation

INTERVENTIONS:
Behavioral: Value-manipulation — During the decision-making task, different choices are assigned different values probabilistically.

SUMMARY:
Learning to make good decisions in the present, and accurately recalling events and information from the past, are critical aspects of human cognition that are often impaired in many psychiatric disorders. This project aims to identify the how the choices individuals make influence what, and how, people remember by combining disparate techniques in computational modeling and direct brain recordings in human subjects. The researcher developed a dual-task paradigm, probing how decisions in one task affect immediate recognition memory. To examine the neural mechanisms underlying model-free RL's influence on memory, the researcher will record local field potential (LFP) and single neuron activity in various brain regions as epilepsy patients perform the proposed task. The results of this project will identify specific neurocomputational mechanisms unifying decision-making and memory processes.

ELIGIBILITY:
Inclusion Criteria:

* Has seizure activity which is deemed non-responsive to standard pharmacological intervention(s), as determined by treating Neurologist and established clinical practices
* Has elected to receive clinically indicated intracranial EEG (electrocorticography (ECoG), stereoelectroencephalography (SEEG)) and/or temporal responsive neurostimulation (RNS) for medication-refractory epilepsy outside of this research study, as determined by treating clinician(s) and per current clinical practice
* Capacity to provide written informed consent
* Language proficiency in English or Spanish
* Willing and able to comply with all study-related procedures

Exclusion Criteria:

* History of psychosis, such as in the context of depressive or manic episode.
* Active suicidal ideation with intent, suicide attempt within the last six months, or other serious suicide risk
* Inability to provide informed consent or reliably participate in study assessments, as per the Montreal Cognitive Assessment (MOCA; score < 26) or in the opinion of the evaluating neuropsychologist.
* Individuals unwilling or unable to undergo electrode implantation procedures
* Medical contraindications to neurosurgery or for general anesthesia, neurosurgery, or an MRI scan (required for electrode implantation)
* Neurological disorder other than epilepsy or other significant brain pathology, if contraindicated in the opinion of implanting neurosurgeon.
* Women who are pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Local-field potentials changes | During task participation, approx. 30-45 min in the first 2 weeks of hospital stay
  Detection of local-field potentials (LFPs) in the various regions (hippocampus, amygdala, and frontal cortex). Local field potentials are the biological voltages recorded by macroelectrodes implanted in participant's subcortical regions as part of their treatment for epilepsy. LFP changes (measured as increases or decreases in voltage) as a function of participant behavior will be recorded, and in response to the task manipulation of the value of choices during the decision-making task
Firing rate changes | During task participation, approx. 30-45 min in the first 2 weeks of hospital stay
  Single-neuron activity recorded from the hippocampus, amygdala, and frontal cortex. Single-neuron activity refers the micro-scale changes in single-neuron action potentials recorded by microelectrodes implanted in subcortical regions. Firing rate changes (measured as difference in spikes/seconds [Hz]) will be reported for neurons as a function of how behavior changes when the value of choices is altered.

SECONDARY OUTCOMES:
Reaction time | During task participation, approx. 30-45 min in the first 2 weeks of hospital stay
  Reaction times involve measuring how quickly the participant makes each choice during the decision-making and memory tasks, in milliseconds. This will be recorded by logging keypresses and mouse inputs to the behavioral computers. Slow reaction times indicate increased cognitive processing.
Number of hit rates for decision-making | During task participation, approx. 30-45 min in the first 2 weeks of hospital stay
  Choices in decision-making task involved logging the decision-making selections that participants make. This will be recorded by logging keypresses and mouse inputs (left or right) to the behavioral computers. This will be used to track whether participants decisions change when value manipulations occur.
Number of hit rates for Memory performance | During task participation, approx. 30-45 min in the first 2 weeks of hospital stay
  Memory performance involved logging the memory-recognition selections that participants make. This will be recorded by logging keypresses and mouse inputs (old or new) to the behavioral computers. This will be used to track whether participants memory performance changes when value manipulations occur.

CONTACTS AND LOCATIONS:
Overall Officials: Salman E Qasim, PhD, Principal Investigator — Icahn School of Medicine at Mt. Sinai
Locations (1):
- Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Access to the raw, de-identified behavioral and neural data will be limited to qualified researchers due to the potential for misuse of participant demographic and neural data within 12 months following article publication. Datasets generated by this project will be made available through the National Institute of Mental Health Data Archive (NDA).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 12 months following article publication
Access Criteria: The datasets will be hosted and available free of charge to approved researchers.